CLINICAL TRIAL: NCT00976547
Title: Correlation Analysis of Hearing Thresholds, Validated Questionnaires and Psychoacoustic Measurements in Tinnitus Patients
Status: Completed | Type: Observational
Sponsor: Faculdade de Medicina de Valenca (Other)
Responsible Party: Ricardo Rodrigues Figueiredo, MD, MSc, OTOSUL, Otorrinolaringologia Sul-Fluminense
Other Study IDs: FMV 2009 001
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2009-09-14 (Estimated); Status verified 2009-09

CONDITIONS: Tinnitus; Hearing Loss; Depression
Keywords: tinnitus; depression; audiometry; measurement
MeSH Terms: conditions — Tinnitus; Hearing Loss; Depression

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tinnitus patients: Group of 48 tinnitus patients

SUMMARY:
Objective: To evaluate the correlation between audiometric thresholds, pitch matching (PM), minimum masking level (MML), Tinnitus Handicap Inventory (THI) and the Beck Depression Inventory (BDI) in tinnitus patients.

Subjects: 48 patients with tinnitus as the main complaint from OTOSUL, Otorrinolaringologia Sul-Fluminense, Volta Redonda, RJ, Brasil and Centro de Tratamento e Pesquisa em Zumbido, Belo Horizonte, MG, Brasil.

Method: Subjects performed tonal audiometry, Pitch Matching (PM) and Minimum Masking Level (MML) for tinnitus. They also fulfilled the Tinnitus Handicap Inventory (THI) and Beck Depression Inventory (BDI). Data was statistically compared for correlation between audiometric thresholds, psycho-acoustic measures and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* tinnitus for more than 6 months
* sensorineural hearing loss
* normal otoscopy

Exclusion Criteria:

* conductive or mixed hearing losses
* A-r, A-d, B and C tympanograms
* tinnitus treatment in the last 6 months
* pregnant woman
* Vestibular Schwannoma

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 48 tinnitus patients sensorineural hearing losses
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo R Figueiredo, MDMSc, Study Chair — OTOSUL, Faculdade de Medicina de Valença
Locations (2):
- Brazil (2):
  - Centro de Diagnóstico e Tratamento do Zumbido, Belo Horizonte, Minas Gerais
  - OTOSUL,Otorrinolaringologia Sul-Fluminense, Volta Redonda, Rio de Janeiro